CLINICAL TRIAL: NCT00400387
Title: Phase III Study Analyzing the Effectiveness of Dalteparin Therapy as Intervention in Recurrent Pregnancy Loss
Brief Title: Effectiveness of Dalteparin Therapy as Intervention in Recurrent Pregnancy Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Ekkehard Schleussner, Sponsor-Investigator, University of Jena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2006-001984-53
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Abortion, Habitual
Keywords: recurrent pregnancy loss
MeSH Terms: conditions — Abortion, Habitual | interventions — Dalteparin; Heparin, Low-Molecular-Weight; levomefolate calcium; Ascorbic Acid; Pyridoxine; Riboflavin; Thiamine; Biotin; Vitamin B 12; Leucovorin

ARMS (2):
- Multivitamin supplement (Other)
  Interventions: Dietary Supplement: Multivitamin supplement
- Multivitamin supplement + dalteparin sodium (Experimental)
  Interventions: Drug: Fragmin P Forte (dalteparin sodium)

INTERVENTIONS:
Drug: Fragmin P Forte (dalteparin sodium) — subcutaneous injection, once daily supported by multivitamine supplement and close monitoring
  Other Names: low molecular weight heparin
  Arms: Multivitamin supplement + dalteparin sodium
Dietary Supplement: Multivitamin supplement — general pregnancy support by multivitamin supplementation and close monitoring
  Other Names: Femibion 800 Folsäure plus Metafolin:; Ascorbinsäure 110 mg; Nicotinamid 15 mg; alpha-Tocopherol acetat 13 mg; RRR-alpha-Tocopherol Äquivalent 7.93 mg; Pantothensäure 6 mg; Pyridoxin 1.9 mg; Riboflavin 1.6 mg; Thiamin 1.2 mg; olsäure 0.4 mg; Biotin 0.06 mg; Cyanocobalamin 0.0035 mg; Calcium mefolinat; Folsäure 0.4 mg; Kalium iodid; Iodid Ion 0.15 mg
  Arms: Multivitamin supplement

SUMMARY:
With this clinical trial the investigators will analyze whether the rate of pregnancy losses before the 24th week of gestation can be reduced by dalteparin treatment in habitual aborters.

DETAILED DESCRIPTION:
Recurrent pregnancy loss (RPL) is a common health problem with three or more loses affecting 1-2% and two or more losses affecting up to 5% of women at the reproductive age (Brenner 2003).

Several aetiologies have been identified or are under discussion to play a role in RPL, including chromosomal translocations and inversions, anatomic alterations of the uterus, endocrinological abnormalities, autoimmune disorders infection, smoking and alcohol consumption, exposure to environmental factors as well as coagulation and immunoregulatory defects (Pandey 2005, Lee 2000). About 30-40% of cases of RPL remain unexplained after standard gynaecological, hormonal and karyotype analysis (Rey 2000).

As stated by Pandey et al (Pandey 2005), a successful implantation during pregnancy requires a balanced equilibrium between coagulation, fibrinolysis and vascular remodeling by the process of angiogenesis in order to avoid excess fibrin accumulation in placental vessels and intervillous spaces (Buchholz 2003). However, thrombosis in decidual vessels is reported to be one of the major causes of RPL (Arias 1998) and could be explained by excessive thrombosis of the placental vessels, placental infarction, and secondary uteroplacental insufficiency.

Recurrent pregnancy loss is a well-described complication of the antiphospholipid antibody syndrome and is thought to be associated with thrombosis of placental vessels, often with evidence for placental infarction. More recently, inherited thrombophilic abnormalities have been linked to RPL and other obstetric complications. At least 16 case-control studies found a high prevalence of factor V Leiden (FVL) in women with unexplained RPL (up to 30%) compared to 1% to 10% of control subjects with odds ratios ranging from 2 to 5 (Press et al. 2002). Likewise, other thrombophilic risk factors including factor II G20210A, hyperhomocysteinemia, protein C, protein S and antithrombin deficiencies have also been associated with RPL (Sanson 1996; Brenner 1999).

A meta-analysis of Rey et al. (Rey 2003) including 31 case control, cohort and cross-sectional studies, showed an association between thrombophilia and fetal loss, though the magnitude varies according to type of fetal loss and type of thrombophilia.

Although most pregnancy losses occur in the first trimester, women with thrombophilia are at an increased risk for pregnancy loss in the second and third trimesters. A number of studies found that FVL carriers have a significantly higher risk of late pregnancy loss than early first trimester loss (Sarig 2002; Meinardi 1999). One possible explanation is that late pregnancy losses may reflect thrombosis of placental vessels. However, the majority of pregnancy losses in women with thrombophilia still occur in the first trimester (Sarig 2002; Younis 2000). The mechanisms responsible for the association of inherited thrombophilia with RPL have not been fully elucidated. Pathological studies of placentas obtained from gestations terminated by foetal loss reveal thrombotic changes and infarcts. These can be observed at the maternal vessels in 50-90% of placentae of women with stillbirth (Gris 1999; Many 2001). However, these changes can also be found in a significant proportion of women with RPL without thrombophilia (Gris 1999; Martinelli 2000). Raising the possibility of yet undetermined gestational prothrombotic risk factors either at fetal vessels or at maternal vessels. A role for foetoplacental thrombosis has been suggested by studies demonstrating an association between factor V genotype in miscarried foetuses and placental infarction. However, the findings of thrombotic changes at the maternal side and the efficacy of LMWH, which do not cross the placentae, in preventing foetal loss are in support with the latter. Emerging data on therapy of women with inherited thrombophilia and pregnancy loss is mostly uncontrolled and include small series of patients treated mainly with LMWH. The potential advantages of LMWH over unfractionated heparin are higher antithrombotic ratio, meaning less bleeding for better antithrombotic effect, longer half-life with a potential need for only one injection per day, smaller injected volume and less heparin-induced thrombocytopenia. These advantages are particularly appealing for prolonged prophylaxis throughout pregnancy and the postpartum period. A recent collaborative study has demonstrated the safety of using LMWH during 486 gestations (Sanson 1999). Successful outcome was reported in 83/93 (89%) gestations in women with recurrent pregnancy loss and in all 28 gestations in women with preeclampsia in previous pregnancy.

Since novel inherited and acquired prothrombotic abnormalities are currently under investigation, clinicians often address the question of prophylaxis in women with RPL who do not have a specific thrombophilic defect. The encouraging results presented above let rise the clinical practise of LMWH therapy without the proved evidence in women without thrombophilic disorders. To give the basis for a rational therapy this question should be answered by this prospective randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy, 5th to 8th week of gestation
* Documented foetal heart activity in US
* History of recurrent pregnancy loss, defined as:

  * 2 or more early (< 12 weeks of gestation) pregnancy losses or
  * 1 or more late (> 12 weeks of gestation) pregnancy loss
* at least 18 years of age
* Written informed consent of the patient

Exclusion Criteria:

* Previous pregnancy losses caused by foetal structural or chromosomal anomalies
* Uterine anomalies
* Maternal infection which caused previous pregnancy loss
* Risk group II or III according to ETHIG I risk stratification (clinical need for heparin prophylaxis)
* Acute thromboembolic event (need of heparin therapy)
* Known hypersensitivity to any of the trial drugs or its ingredients (i.e. thrombocytopenia type II caused by allergic reaction to heparin)
* Antiphospholipid antibody syndrome
* Diabetes mellitus
* Ongoing nicotine or drug or alcohol abuse
* Known HIV infection
* Expected low compliance (e.g. by travel distance to trial site)
* Current or recent (within 30 days prior to start of trial treatment) treatment with another investigational drug or participation in another investigational trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2006-11; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
ongoing intact pregnancy at 24 weeks of gestation | at 24 weeks of gestation

SECONDARY OUTCOMES:
late pregnancy complication, defined as at least one of the following: preterm delivery, placenta insufficiency, intrauterine growth retardation, preeclampsia and abruptio placentae | 6-8 weeks after delivery
foetus with structural anomalies | 6-8 weeks after delivery
side effects of dalteparin therapy (e.g. thrombocytopenia, osteoporosis, haemorrhage) | 6-8 weeks after delivery
life birth | 6-8 weeks after delivery
preterm delivery (< 37 weeks of gestation) | 6-8 weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Schleussner, Prof. Dr., Principal Investigator — University of Jena, Hospital for gynaecology and obstetrics
Locations (12):
- Kinderwunschinstitut Schenk, Dobl, Austria
- Germany (11):
  - Martin-Luther-Universität Halle Wittenberg, Halle, Saxony-Anhalt
  - Universitätsfrauenklinik am Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - Krankenhaus St. Elisabeth und St. Barbara, Klinik für Frauenheilkunde und Geburtshilfe, Halle
  - Medizinische Hochschule Hannover, Abt. für Gynäkologie und Geburtshilfe, Hanover
  - Frauenklinik Landshut Achdorf, Landshut
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Klinikum der Universität München Großhadern, Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, München
  - Frauenklinik der Technischen Universität München, Klinikum rechts der Isa, München
  - Praxis für medizinische Genetik, Regensburg
  - Klinikum Stuttgart, Frauenklinik, Stuttgart
  - Universitätsfrauenklinik Tübingen, Tübingen

REFERENCES:
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986
- [Derived] Rogenhofer N, Markoff A, Wagner A, Klein HG, Petroff D, Schleussner E; EThIG II Group; Thaler CJ. Lessons From the EThIGII Trial: Proper Putative Benefit Assessment of Low-Molecular-Weight Heparin Treatment in M2/ANXA5 Haplotype Carriers. Clin Appl Thromb Hemost. 2017 Jan;23(1):27-33. doi: 10.1177/1076029616658117. Epub 2016 Jul 14. PMID 27418639
- [Derived] Schleussner E, Kamin G, Seliger G, Rogenhofer N, Ebner S, Toth B, Schenk M, Henes M, Bohlmann MK, Fischer T, Brosteanu O, Bauersachs R, Petroff D; ETHIG II group. Low-molecular-weight heparin for women with unexplained recurrent pregnancy loss: a multicenter trial with a minimization randomization scheme. Ann Intern Med. 2015 May 5;162(9):601-9. doi: 10.7326/M14-2062. PMID 25938990
- See also: Related Info — http://www.geburtshilfe.uniklinikum-jena.de/ETHIG_II__Studie.html